CLINICAL TRIAL: NCT02788240
Title: To Study the Influence of GCSF on Natural History of Acute On Chronic Liver Failure After the Acute Phase - A Randomized Controlled Study
Brief Title: To Study the Influence of GCSF on Natural History of Acute On Chronic Liver Failure After the Acute Phase
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-ACLF-008
Record Dates: First submitted 2016-03-22; First posted 2016-06-02 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Albumins; Nutritional Status; Terlipressin; Meropenem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peg GCSF with standard medical therapy (Experimental)
  Interventions: Drug: Peg GCSF; Biological: 20% Albumin; Dietary Supplement: Nutrition; Other: Bowel wash; Drug: Terlipressin 1- 4mg,if indicated; Drug: Meropenem or Imepenem, if indicated
- Placebo with standard medical therapy (Active Comparator)
  Interventions: Biological: 20% Albumin; Dietary Supplement: Nutrition; Other: Bowel wash; Drug: Terlipressin 1- 4mg,if indicated; Drug: Meropenem or Imepenem, if indicated; Drug: Placebo

INTERVENTIONS:
Drug: Peg GCSF
  Arms: Peg GCSF with standard medical therapy
Biological: 20% Albumin
Dietary Supplement: Nutrition
Other: Bowel wash
Drug: Terlipressin 1- 4mg,if indicated
Drug: Meropenem or Imepenem, if indicated
Drug: Placebo
  Arms: Placebo with standard medical therapy

SUMMARY:
All consecutive ACLF (Acute on Chronic Liver failure) patients presenting to the institute of liver and biliary sciences, irrespective of the etiology , who have survived the acute phase (i.e. 90 days of onset of the acute on chronic liver failure) and who are willing to participate in the study would be enrolled. After performing baseline biochemical tests, patients will undergo transjugular liver biopsy (TJLB), HVPG (Hepatic Venous Pressure Gradient), Circulating CD34 cells, Bone marrow aspiration and biopsy (Histopathological and immunohistochemical examination will be done).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65 years
* All patients who were known to have ACLF and have survived 3 months of the onset of acute event
* Patients willing to participate in the study

Exclusion Criteria:

* Presence of AKI (Acute Kidney Injury)
* Active sepsis (Blood/ urine culture positive, SBP (Spontaneous bacterial Peritonitis, LRTI (lower Respiratory Tract infection)
* Sickle cell anemia
* HepatoCellular Carcinoma
* Hematological malignancies
* Multi organ failure
* Grade 3/ 4 HE (Hepatic Encephalopathy)
* HIV seropositivity
* Pregnancy
* Patients being taken up for transplant
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Transplant free survival in both groups | 1 year

SECONDARY OUTCOMES:
Quantitative assessment of CD34 positive cells in serum in both groups. | 1 year
  On Immunohistochemistry of liver biopsy tissue,quantification of + ve CD34 cells will be done
Quantitative assessment of CD34 positive cells in liver biopsy samples in both groups. | 1 year
  On Immunohistochemistry of liver biopsy tissue,quantification of + ve CD34 cells will be done
Reduction in liver disease severity indices like CTP (Child-Turcotte-Pugh) by more than one point in both groups. | 1 year
Reduction in liver disease severity indices like MELD Na ((Model for End Stage liver disease) by more than 2 points in both groups. | 1 year
Development of new onset complications such as hepatic encephalopathy in both groups. | 1 year
Development of new onset complications such as hepatorenal syndrome in both groups. | 1 year
Development of new onset complications such as sepsis in both groups. | 1 year
Development of new onset complications such as Hepatocellular carcinoma (HCC). | 1 year
Total number of CD34 positive cells in histopathological examination of bone marrow in both groups | 1 year
No of adverse events in both groups | 1 year
Reduction in HVPG (Hepatic Venous Pressure Gradient) in both groups | 1 year
Reduction in HBV DNA level in both groups. | 1 year
Number of patients who will restart alcohol abuse during the follow up period in both groups. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No